CLINICAL TRIAL: NCT02735694
Title: Cycloserine in the Treatment of Sleep Apnea
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Analysis of initial sample shows negative results.
Sponsor: University of Manitoba (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B2013:044; MA-7954 (Other Grant/Funding Number: CIHR); 9427-U0304-36C (Other: Health Canada)
Record Dates: First submitted 2015-11-18; First posted 2016-04-13 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2015-11

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep apnea; Hypoglossal Nerve; N-methyl-D-aspartate receptors; Cycloserine; Short-term potentiation
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Cycloserine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cycloserine (Active Comparator): Cycloserine, 250 mg capsules by mouth, one hour prior to initiation of sleep study, single dose
  Interventions: Drug: Cycloserine; Drug: Placebo
- Placebo (Placebo Comparator): Placebo, sugar capsule by mouth, one hour prior to initiation of sleep study, single dose
  Interventions: Drug: Cycloserine; Drug: Placebo

INTERVENTIONS:
Drug: Cycloserine — Capsule containing 250 mg of Cycloserine
  Other Names: Seromycin
Drug: Placebo — Sugar capsule manufactured to mimic Cycloserine 250 mg capsule
  Other Names: Sugar capsule

SUMMARY:
This study is being conducted to determine whether cycloserine is effective for the treatment of sleep apnea. Cycloserine is an antibiotic that has been extensively used in the treatment tuberculosis. However, more recently it was shown to enhance memory responses. Cycloserine may enhance the response of respiratory muscles to apnea and potentially reduce the severity of sleep disordered breathing.

DETAILED DESCRIPTION:
The passive human upper airway (UA) is a collapsible tube with a relatively high compliance. At atmospheric luminal pressure, its cross-sectional area varies considerably. Subjects in whom the pharynx is closed, or nearly closed, at near atmospheric pressure require an upper airway dilating force to maintain adequate ventilation. During wakefulness pharyngeal dilator muscles (dilators) provide the necessary force to permit an adequate flow, regardless of how collapsible the pharynx is. This dilator activity is substantially lost at sleep onset. Subjects in whom the passive UA cannot permit adequate ventilation must recruit dilators through reflex mechanisms if they are to remain asleep. Recent studies have shown that activation of the muscles that open the airway in the course of obstructive apneas persists to a variable degree after the relief of obstruction, evidencing the presence of memory for prior activation in the the brain centers that supply the dilator muscles.

Short-term potentiation (STP) is a neuro-physiological mechanism that results in a time-dependent increase in motor activity, that is not explainable by changes in stimulus intensity, and which persists after disappearance of the stimulus ( "after-discharge"). STP is well documented in diaphragmatic responses to chemical stimuli. Prominent STP in upper airway muscles would promote a stronger dilator response to upper airway occlusion. The after-discharge would also help to maintain dilator activity following the ventilatory phase of obstructive events, thereby mitigating recurrence of obstruction. Patients with obstructive sleep apnea (OSA) vary greatly in the extent to which this memory or STP is present. The investigators postulate that interventions that could potentiate the development of memory for prior activation would mitigate the recurrence of apneas and reduce the severity of obstructive sleep apnea. The same interventions, those that enhance memory for prior activation, would also likely improve central apneas in that these apneas represent loss of diaphragm activity following hyperventilation. Memory for prior activation of the diaphragm has been well documented in the past and appears to be defective in such patients.

There has been extensive research into methods of improving neural memory. Cycloserine, an antibiotic that has been, and continues to be, used extensively in the treatment of drug-resistant tuberculosis, was shown to be effective in promoting memory in small doses (much less than those used for tuberculosis) both in animals and humans. We, therefore, propose that cycloserine has the potential of enhancing the memory properties of neurones supplying pharyngeal muscles and propose to study the effect of using it on the severity of sleep apneas of the obstructive and central varieties.

Patients who have been diagnosed with OSA following routine clinical sleep studies will be asked to participate. Participation involves agreeing to two additional full night studies in the sleep laboratory, separated by 1 week. Both studies will be identical to the routine clinical studies, except that the patient will be asked to swallow a capsule containing either placebo or 250 mg cycloserine 1 to 2 hours prior to going to sleep. The order of the Placebo and Test nights will be randomized. The patient will be monitored continuously by a dedicated, senior polysomnography technologist.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe obstructive or central sleep apnea (Apnea Hypopnea Index > 30/hr).
* Minimum Oxygen saturation during respiratory events >70% throughout sleep during the clinical sleep study.

Exclusion Criteria:

* Contraindication to the use of cycloserine, namely history of allergy to cycloserine, seizures, depression, severe anxiety or psychosis, excessive use of alcohol or renal failure.
* Past or current history of tuberculosis
* Hypercapnia > 55 millimeters of mercury during the diagnostic clinical sleep study.
* Neuromuscular disease.
* Obesity-hypoventilation syndrome.
* Pregnancy.
* Significant co-morbidities: Dialysis-dependant renal failure, severe asthma or chronic lung disease, congestive heart failure, previous stroke.
* Recent (within 3 months) myocardial infarction or Active coronary ischemia event.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Apnea-hypopnea index (AHI) | Baseline and one week
  Baseline apnea-hypopnea index in first night and upon end of the second sleep study, performed one week apart

SECONDARY OUTCOMES:
Improvement in total sleep time | Baseline and one week
Improvement in average oxygen saturation | One week

OTHER OUTCOMES:
Improvement in the awakening and arousals index | One week
  number of awakenings and arousals per hour of sleep as measurement of sleep continuity.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy K Younes, Md, PhD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Sleep Disorders Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No
No plan has been made on sharing individual data